CLINICAL TRIAL: NCT02110563
Title: Phase I, Multicenter, Cohort Dose Escalation Trial to Determine the Safety, Tolerance, and Maximum Tolerated Dose of DCR-MYC, a Lipid Nanoparticle (LNP)-Formulated Small Inhibitory RNA (siRNA) Oligonucleotide Targeting MYC, in Patients With Refractory Locally Advanced or Metastatic Solid Tumor Malignancies, Multiple Myeloma, or Lymphoma
Brief Title: Phase I, Multicenter, Dose Escalation Study of DCR-MYC in Patients With Solid Tumors, Multiple Myeloma, or Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCR-MYC-101
Record Dates: First submitted 2014-04-06; First posted 2014-04-10 (Estimated); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Solid Tumors; Multiple Myeloma; Non-Hodgkins Lymphoma; Pancreatic Neuroendocrine Tumors; PNET; NHL
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Neuroectodermal Tumors, Primitive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DCR-MYC (Experimental): Patient groups (cohorts) will receive a single dose level of DCR-MYC; the dose level of DCR-MYC will be increased in subsequent cohorts
  Interventions: Drug: DCR-MYC

INTERVENTIONS:
Drug: DCR-MYC — Dosing: 2 hour IV infusion on Day 1 and 8 of each 21 day cycle.
  Starting dose: 0.1mg/kg/dose
  Dose escalation: 100%, 50%, or 25% increase in subsequent cohorts depending upon toxicity.
  Number of cycles: until progression or unacceptable toxicity develops.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of the investigational anticancer drug DCR-MYC. DCR-MYC is a novel synthetic double-stranded RNA in a stable lipid particle suspension that targets the oncogene MYC. MYC oncogene activation is important to the growth of many hematologic and solid tumor malignancies. In this study the Sponsor proposes to study DCR-MYC and its ability to inhibit MYC and thereby inhibit cancer cell growth.

DETAILED DESCRIPTION:
In this first-in human study, DCR-MYC will be administered by 2 hour intravenous (IV) infusion, once weekly for 2 weeks followed by a rest week (3 weeks = 1 cycle), to patients with either solid tumor malignancies, multiple myeloma, or non-Hodgkins lymphoma that have not responded to previous treatment. The highest safe dose of DCR-MYC that can be administered will be identified. In addition, the pharmacokinetic (PK) profile, potential pharmacodynamic (PD) effects, as well as the antitumor activity of DCR-MYC will be evaluated.

There will be 2 expansion cohorts at the maximum tolerated dose (MTD) (or highest safe dose identified for further study which may be lower):

* Biopsy Cohort: 6 patients, tumor biopsies to be performed pre-dosing and Cycle 2/Day 11; same assessments as dose escalation cohorts
* PNET Cohort: Up to 20 patients with pancreatic neuroendocrine tumors; same assessments as dose escalation cohorts, however fewer PD (cytokine) assessments and no PK assessments

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, > 18 years of age at the time of obtaining informed consent.
2. Patients with a documented solid tumor malignancy that is locally advanced or metastatic; patients with documented multiple myeloma or non-Hodgkin's lymphoma.
3. Patients with a malignancy that is either refractory to standard therapy or for which no standard therapy is available.
4. Patients with a malignancy that is currently not amenable to surgical intervention due to either medical contraindications or non-resectability of the tumor.
5. Dose escalation portion of study: Patients with measurable or non-measurable disease according to standard response criteria .
6. MTD Biopsy Cohort ONLY: Patients with measurable disease with primary or metastatic tumor site(s) considered safely accessible for biopsy; patients must consent to undergo 2 tumor biopsies.
7. MTD PNET Cohort ONLY: Patients with advanced (unresectable or metastatic), histologically-confirmed low or intermediate grade PNET according to the World Health Organization (WHO) 2010 classification. Patients with neuroendocrine tumors (e.g., gastrinoma, VIPoma) in whom a pancreatic or peripancreatic primary is strongly suspected are also eligible. Patients must also have:

   * A Ki-67 proliferation index < 20%
   * Demonstrated radiological evidence of disease progression during or following the last treatment regimen (based on CT, MRI, or Octreoscan®)
   * Measurable disease according to RECIST v1.1 (determined by CT or MRI). Any lesions which have been subjected to percutaneous therapies or radiotherapy should not be considered measureable, unless the lesion has clearly progressed (per RECIST v1.1) since the procedure.
   * Received < 2 prior systemic treatments for PNET, at least one of which must have been an FDA-approved targeted therapy for PNET (i.e., sunitinib [Sutent®] or everolimus [Afinitor®]). Treatment with a somatostatin analog (SSA) will not be considered as a systemic treatment for the purposes of eligibility.
8. Patients with an Eastern Cooperative Oncology Group performance status of 0, 1, or 2, and an anticipated life expectancy of ≥ 3 months.
9. Patients, both male and female, who are either not of childbearing potential or who agree to use a medically effective method of contraception during the study and for 3 months after the last dose of study drug.
10. Patients with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol.

Exclusion Criteria-Patients:

1. Women who are pregnant or lactating. Women of child-bearing potential (WOCBP), and fertile men with a WOCBP-partner not using and not willing to use a medically effective method of contraception.
2. Patients with known central nervous system (CNS) or leptomeningeal metastases not controlled by prior surgery or radiotherapy, or patients with symptoms suggesting CNS involvement for which treatment is required.
3. Patients with leukemia (any form) or myelodysplastic syndromes.
4. MTD PNET Cohort ONLY: Patients with poorly differentiated, high grade (grade 3) neuroendocrine carcinoma, as well as patients with adenocarcinoid, goblet cell carcinoid, or small cell carcinoma, or PNET patients with a Ki-67 proliferation index > 20 %.
5. Patients with any of the following hematologic abnormalities at baseline:

   * Absolute neutrophil count < 1,500 per mm3
   * Platelet count < 100,000 per mm3
6. Patients with any of the following serum chemistry abnormalities at baseline:

   * Total bilirubin > 1.5 × the ULN for the institution
   * AST or ALT > 3 × the ULN for the institution (> 5 × if due to hepatic involvement by tumor)
   * Creatinine > 1.5 × ULN for the institution
7. Patients with any of the following coagulation parameter abnormalities at baseline:

   * PT (INR) > 1.5 × ULN for the institution
   * PTT > 1.5 × ULN for the institution
8. Patients with:

   * Active thrombosis, or a history of deep vein thrombosis or pulmonary embolism, within 6 months prior to first study drug administration; patients receiving systemic anti-coagulation for prophylactic or therapeutic reasons
   * Active uncontrolled bleeding or a known bleeding diathesis
9. Patients with a significant cardiovascular disease or condition, including:

   * Congestive heart failure currently requiring therapy
   * Need for antiarrhythmic medical therapy for a ventricular arrhythmia
   * Severe conduction disturbance (e.g., 3rd degree heart block)
   * Angina pectoris requiring therapy
   * Known left ventricular ejection fraction < 50% by MUGA or echocardiogram
   * QTc interval > 450 msec in males, or > 470 msec in females
   * Uncontrolled hypertension (per the Investigator's discretion)
   * Class III or IV cardiovascular disease according to the New York Heart Association's Functional Criteria.
   * Myocardial infarction within 6 months prior to first study drug administration
10. Patients with a known or suspected hypersensitivity to any of the components of lipid nanoparticle-formulated DCR-MYC.
11. Patients with a known history of human immunodeficiency virus or active infection with hepatitis B virus or hepatitis C virus.
12. Patients with any other serious/active/uncontrolled infection, any infection requiring parenteral antibiotics, or unexplained fever > 38ºC within 2 weeks prior to first study drug administration.
13. Patients with inadequate recovery from an acute toxicity associated with any prior antineoplastic therapy.
14. Patients with inadequate recovery from any prior surgical procedure, or patients having undergone any major surgical procedure within 4 weeks prior to first study drug administration.
15. Patients with any other life-threatening illness, significant organ system dysfunction, or clinically significant laboratory abnormality, which, in the opinion of the Investigator, would either compromise the patient's safety or interfere with evaluation of the safety of the study drug.
16. Patients with a psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary study-related evaluations.
17. Patients with the inability or with foreseeable incapacity, in the opinion of the Investigator, to comply with the protocol requirements.

Exclusion Criteria-Treatments:

1. MTD PNET Cohort ONLY: Greater than 2 prior systemic treatments for the underlying malignancy
2. Any antineoplastic agent for the primary malignancy (standard or experimental) within 4 weeks prior to first study drug administration with the exception of monoclonal antibody therapy, nitrosoureas, and nitrogen mustard for the primary malignancy within 6 weeks prior to first study drug administration
3. Radiotherapy for the primary malignancy within 4 weeks prior to first study drug administration and during study.
4. Herbal preparations or related over-the-counter preparations/supplements containing herbal ingredients within 2 weeks prior to first study drug administration and during study.
5. Systemic hormonal therapy within 2 weeks prior to first study drug administration and during study.
6. Any other investigational treatments during study. This includes participation in any medical device or therapeutic intervention clinical trials.
7. Prophylactic use of hematopoietic growth factors within 1 week prior to first study drug administration and during Cycle 1 of study; thereafter prophylactic use of growth factors is allowed as clinically indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2016-11-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | Cycle 1 (3 weeks), longer if DRC-MYC is continued; with 30 days follow-up after last dose
  Part A: 1 patient cohorts with 100% dose increase between cohorts until >/= Grade 2 study drug-related toxicity during Cycle 1, then expand to 3 patients and move to Part B.
  Part B: 3 patient cohorts with 50% dose increase between cohorts until study drug-related DLT during Cycle 1, then expand to 6 patients and move to Part C.
  Part C: 3 to 6 patient cohorts with 25% dose increase between cohorts until > 1 study drug-related DLT, then stop escalation and expand previous MTD cohort to 18 patients.

SECONDARY OUTCOMES:
DCR-MYC levels in blood | Cycle 1; Week 1 and Week 2
  Samples to be collected Week 1 (Day 1, 2, and 4) and Week 2 (Day 8 and 11)
DCR-MYC biological activities | Cycle 1; Week 1 and Week 2
  Collection of blood samples for cytokine measurements Week 1 (Day 1, 2, and 4) and Week 2 (Day 8)
DCR-MYC biological activities | Cycle 1, Cycle 2, and Cycle 4
  PET imaging to be performed Cycle 1/Day 1, Cycle 1/Day 11, and End of Cycle 4
DCR-MYC biological activities | Cycle 1 and Cycle 2
  Tumor biopsies (2 total) to be performed in MTD expansion cohort only. Patients will have biopsies performed prior to Cycle 1 and Cycle 2/Day 11
Preliminary antitumor activity | After Cycle 2 (6 weeks), then at 6 week intervals if DCR-MYC is continued
  Evaluation for evidence of objective response or disease stabilization

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Stanford Cancer Institute, Stanford, California
  - University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - South Texas Accelerated Research Therapeutics (START)-Midwest, Grand Rapids, Michigan
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No